CLINICAL TRIAL: NCT07121647
Title: Selective Plasmofiltration in the Treatment of Patients With Abdominal Septic Shock: a Prospective Interventional Controlled Study
Brief Title: Selective Plasmofiltration for Abdominal Septic Shock: a Clinical Ctudy
Acronym: SPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Masolitin Sergey Viktorovich, Assistant Professor of Anesthesiology and Critical Care, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 31_05_2016_№5; 31.05.2016.5.Pirogov (Other: 31.05.2016.5.Pirogov)
Record Dates: First submitted 2025-03-10; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Selective Plasma Filtration
Keywords: septic shock; interleukin-6; continuous renal replacement therapy; selective plasmofiltration,
MeSH Terms: conditions — Shock, Septic | interventions — Renal Replacement Therapy

STUDY DESIGN:
Intervention Model Description: Patients who showed no clinical improvement within 12 hours of admission to the intensive care unit (ICU) (pH ≤ 7.2, lactate ≥ 2.0 mmol/L, base deficit ≤ -2.0 mmol/L) were randomized using a random number generator and divided into three groups:
  Group 1 (n=34): Patients received standard conservative therapy combined with isolated prolonged veno-venous hemodiafiltration (CVVHDF), which was initiated upon the occurrence of urgent indications for renal replacement therapy (RRT), such as uremia, oliguria, and hyperkalemia.
  Group 2 (n=35): Patients underwent early isolated CVVHDF.
  Group 3 (n=32): Patients received early combined extracorporeal blood purification therapy (EBPT) (SPF and CVVHDF).
Masking Description: The first stage involved standard clinical and laboratory monitoring, along with daily assessment of the severity of the patients' condition.
  The second stage included the distribution of patients into three groups. The third stage involved the implementation of renal replacement therapy (RRT). The fourth stage consisted of statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (n=34) (Other): Patients got standard conservative therapy in accordance with the principles of the survive sepsis compain (SSC) in combination with isolated continuous veno-venous hemodiafiltration (cvvhdf), which started in the presence of absolute indications such as acidemia, hyperhydration with pulmonary edema, hyperkalemia).
  Interventions: Procedure: renal replacement therapy.
- Group 2 (n=35) (Active Comparator): Patients got standard conservative therapy accordingly with SSC in combination with early isolated veno-venous hemodiafiltration started with AKI 1 stage KDIGO.
  Interventions: Procedure: early isolated CVVHDF.
- Group 3 (n=32) (Experimental): Patients got standard conservative therapy in accordance with SSC in combination with extracorporeal blood purification therapies (EBPT) including a selective plasmafiltration in combination with cvvhdf.
  Interventions: Procedure: combined extracorporeal blood purification therapy

INTERVENTIONS:
Procedure: renal replacement therapy. — veno-venous hemodiafiltration for emergency indications (CVVHDF).
  Arms: Group 1 (n=34)
Procedure: early isolated CVVHDF. — early isolated CVVHDF.
  Arms: Group 2 (n=35)
Procedure: combined extracorporeal blood purification therapy — Patients received early combined extracorporeal blood purification therapy (EBPT) (SPF and CVVHDF).
  Arms: Group 3 (n=32)

SUMMARY:
Group 1: 34 patients received prolonged hemodiafiltration (CVVHDF) on an emergency basis.

Group 2: 35 patients received early isolated CVVHDF. Group 3: 32 patients received early combined extracorporeal detoxification (ECD) (selective plasma filtration [SPF] + CVVHDF).

A comparative analysis of clinical and laboratory parameters was performed.

DETAILED DESCRIPTION:
Prospective Single-Center Interventional Study Conducted at City Clinical Hospital No. 1 Named After N.I. Pirogov, Including 101 Patients with Abdominal Septic Shock Complicated by Acute Kidney Injury

The study was approved by the Ethics Committee of the hospital (Protocol No. 7, dated May 31, 2016).

Inclusion Criteria: Simultaneous presence of clinical and laboratory signs of septic shock, as defined by the Sepsis-3 criteria , and clinical presentation of acute kidney injury corresponding to Stage 1 of the KDIGO classification:

Severity of organ dysfunction assessed by the SOFA (Sepsis-related Organ Failure Assessment) score > 2 points, as a result of a confirmed or suspected infection focus;

The need for vasopressors to maintain a mean arterial pressure ≥65 mmHg and a serum lactate level >2 mmol/L after adequate fluid resuscitation.

Exclusion Criteria: Terminal condition, ongoing internal bleeding, atonic coma, severe heart failure (left ventricular ejection fraction <25%), decompensated liver failure, body weight less than 20 kg, age <18 years, pregnant women, septic shock without acute kidney injury.

Exclusion from the Study: Patient refusal to continue participation; deviations from the study protocol.

Study Limitation: Limited availability of consumables (plasma separators) during the study period.

The study was structured into six consecutive stages:

Stage I - Clinical and Laboratory Monitoring and Scoring of Patients: Standard monitoring of hemodynamic and clinical-laboratory parameters was performed. For statistical analysis, the worst parameter recorded within 24 hours was considered. The SOFA score (daily), APACHE II score (on admission), and KDIGO classification for acute kidney injury were used to assess organ dysfunction severity. Glomerular filtration rate (GFR) was estimated using the CKD-EPI 2021 formula (Chronic Kidney Disease Epidemiology Collaboration) based on serum cystatin-C levels. Concentrations of cytokines (interleukin-6 [IL-6], tumor necrosis factor [TNF]), and low- and middle-molecular-weight substances (LMMWS) in serum were measured on days 1 (before the procedure), 2, 3, 5, 7, and 10 of therapy.

Stage II - Comprehensive Intensive Therapy: Conducted in accordance with international guidelines for the management of sepsis and septic shock.

Stage III - Patient Group Allocation: Patients who, within 12 hours of admission to the ICU and surgical source control, could not achieve correction of acid-base balance (pH ≤ 7.2, lactate ≥ 2.0, BE ≤ -2.0) despite escalating doses of vasopressors and persistent acute kidney injury, were randomized into groups based on the timing and modality of extracorporeal detoxification (ECD). Randomization was performed using the Jamovi software (version 2.6.24) with the built-in R function. Three columns were created: the first for patient IDs (1 to 105), the second for group numbers (1 to 3), and the third for the R code: sample(rep(1:3, each = 35)). This code generated a vector with numbers from 1 to 3 (each number repeated 35 times) and shuffled them randomly. The results were exported to Excel.

Group 1: 34 patients continued to receive conservative intensive therapy until classical indications for renal replacement therapy (RRT) emerged, such as severe kidney dysfunction posing an immediate threat to life (uremia with blood urea >40 mmol/L; anuria or oliguria refractory to diuretics; serum potassium >6.5 mmol/L). RRT was performed as delayed isolated prolonged veno-venous hemodiafiltration (PVVHDF).

Group 2: 35 patients received early isolated PVVHDF in addition to standard intensive therapy.

Group 3: 32 patients received selective plasma filtration (SPF) before early isolated PVVHDF. Each patient underwent 4 SPF procedures (on days 1, 2, 3, and 5).

Stage IV - ECD Procedures: PVVHDF for all groups was performed in post-dilution mode (multiFiltrate: Fresenius Medical Care) using the "Kit-8" cartridge and AV1000S hemofilter (surface area = 1.8 m²). Blood flow rate was 150-200 mL/min. The dose of renal replacement therapy was 30-40 mL/kg/day (total effluent and ultrafiltrate volume relative to patient body weight). Ultrafiltration volume and rate were adjusted individually. PVVHDF duration ranged from 24 to 72 hours. Systemic anticoagulation was achieved with bolus unfractionated heparin: 30-50 IU/kg at the start, followed by 10-20 IU/kg/hour (500-1000 IU/hour), monitored by activated partial thromboplastin time (aPTT). SPF was performed using EVACLIO-EC-2C20 plasma separators (Kawasumi, Japan) in membrane plasma separation mode (multiFiltrate: Fresenius Medical Care). Perfusion rate was 120 mL/min. Plasma replacement during SPF was performed with 20% albumin solution (200 mL) in an isovolemic solution (ACCUSOL 4 K+ 5000 mL). Replacement volume ranged from 2 to 3 times the circulating plasma volume (5-10 liters). Anticoagulation: unfractionated heparin 2000 IU/hour (into the arterial segment of the circuit before the plasma separator).

Stage V - Dynamic Clinical and Laboratory Monitoring: Conducted on days 1, 2, 3, 5, 7, and 10 in the ICU.

Stage VI - Statistical Analysis: Data are presented as median and interquartile range (25th and 75th percentiles). The Kolmogorov-Smirnov test was used to assess data normality. Non-parametric Mann-Whitney U test was used for intergroup comparisons. The Wilcoxon signed-rank test was used to assess changes over time. Fisher's exact test was used for qualitative data. Logistic regression was used to assess posterior probabilities. Survival analysis was performed using the Kaplan-Meier method. Spearman's rank correlation was used to assess correlations. A p-value <0.05 was considered statistically significant. Data analysis was performed using SPSS-27.0 and Jamovi-2.6.2024 software.

ELIGIBILITY:
Inclusion Criteria:

Abdominal septic shock (Sepsis-3) and AKI stage 1 according to the KDIGO (Kidney Disease Improving Global Outcomes) classification

Exclusion Criteria:

Terminal state, active bleeding, atonic coma, severe heart failure (left ventricular ejection fraction <25%), decompensated liver failure, body weight less than 20 kg, age under 18 years, pregnancy, as well as cases of septic shock without AKI.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
analysis of hospital mortality | hospital mortality from the moment of randomization (point 0) and then on 2,4,6,8,10,12,14 and 30 days
  Estimation of hospital mortality is by means Fisher's exact test.
length of stay in the ICU | The duration of staying in the ICU, measured from the moment of randomization (point 0) and then until the moment of transfer to the specialized department on 2,4,6,8,10,12,14 and 30 days
  Length of stay in the ICU was evaluated.
Length of hospital stay | differences in the duration of hospitalization measured from the moment of randomization (point 0) and then on 2,4,6,8,10,12,14 and 30 days in days of staying in the clinic
  Time from arriving to leaving hospital was estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov Russian National Research Medical University (RNRMU),, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the findings of this study will be openly available in the Figshare repository.
Supporting Information: SAP, CSR
Time Frame: 10.03.2025
Access Criteria: Open access
URL: https://doi.org/10.6084/m9.figshare.28512992

REFERENCES:
- See also: Blood purification in abdominal septic shock with acute kidney injury: a prospective interventional controlled study (part I) — https://doi.org/10.6084/m9.figshare.28512992
- See also: Blood purification in abdominal septic shock with acute kidney injury: a prospective interventional controlled study (part II) — https://doi.org/10.6084/m9.figshare.28513046